CLINICAL TRIAL: NCT02451033
Title: Granulocyte Colony Stimulating Factor And Growth Hormone In Cirrhosis Of Liver: An Open Label Study
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Dr.Virendra Singh, Professor of Hepatology, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: G-CSF and GH in cirrhosis
Record Dates: First submitted 2015-05-12; First posted 2015-05-21 (Estimated); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Cirrhosis
Keywords: Regenerative medicine
MeSH Terms: conditions — Fibrosis | interventions — Granulocyte Colony-Stimulating Factor; Growth Hormone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- standard medical therapy (Active Comparator): Standard medical therapy
  Interventions: Drug: standard medical therapy
- G-CSF (Active Comparator): Standard medical therapy plus G-CSF at the dosage of 5 µg/Kg subcutaneously every 12 hr for five consecutive days then every 3 monthly for 3 days till 1 year.
  Interventions: Drug: standard medical therapy; Drug: G-CSF
- G-CSF plus growth hormone (Active Comparator): Standard medical therapy plus G-CSF plus Growth Hormone therapy. Growth Hormone will be given in low dose of 1unit sc daily for 1 year.
  Interventions: Drug: standard medical therapy; Drug: G-CSF; Drug: Growth Hormone

INTERVENTIONS:
Drug: standard medical therapy — diuretics, albumin infusion, antibiotics, nutrition, and variceal banding wherever needed
Drug: G-CSF — G-CSF at the dosage of 5 µg/Kg subcutaneously every 12 hr for five consecutive days then every 3 monthly for 3 days till 1 year
  Arms: G-CSF; G-CSF plus growth hormone
Drug: Growth Hormone — Growth Hormone in low dose of 1unit sc daily for 1 year
  Arms: G-CSF plus growth hormone

SUMMARY:
Cirrhosis of liver is a leading cause of morbidity and mortality worldwide . Complications including ascites, spontaneous bacterial peritonitis (SBP), variceal bleed, hepatic encephalopathy, hepatorenal syndrome (HRS) and development of hepatocellular carcinoma (HCC) have poor prognosis and further decreases the survival in these patients. It has been believed that cirrhosis is irreversible and that treatment should focus on preventing the progression of liver fibrosis/dysfunction and its complications.

Currently the only effective treatment is liver transplantation, an increasingly limited and expensive resource especially in developing countries. Furthermore, transplantation comes with a requirement for lifelong immunosuppression, and considerable long-term side effects that include chronic renal failure, post-transplant lymphoproliferative disease, and cardiovascular complications.

Short of liver transplant, recently, reports of unexpected plasticity in adult bone marrow have raised hopes that stem cell therapy may offer exciting therapeutic possibilities for patients with end stage liver diseases. It has been shown that in response to acute or chronic liver damage, bone marrow derived stem cells can spontaneously populate the liver and differentiate into hepatic cells. Animal and human studies suggested that such cells might contribute to the regeneration after different kinds of liver injuries . In animal models, after liver injury, bone marrow-derived circulating pluripotent cells have been reported to participate in liver repopulation with both non-parenchymal cells and hepatocytes. This repopulation process, however, seems to be highly dependent on the type of liver injury and experimental conditions. Fusion with hematopoietic cells has been substantiated as a mechanism by which hepatocytes can regenerate, and studies have demonstrated improved liver histology and survival in patients with cirrhosis following mobilization of bone marrow stem cells by granulocyte-colony stimulating factor (G-CSF) . Three recent studies have demonstrated G-CSF induced mobilization of bone marrow stem cells (CD34 cells) in peripheral blood and their subsequent increase in liver tissue and improved survival in patients with alcoholic hepatitis and acute on chronic liver failure (ACLF) . However there is insufficient data on whether G-CSF improves survival and prognosis in patients with cirrhosis.

Also, Malnutrition is commonly seen (60-70%) in cirrhotics and have adverse prognosis on its outcome . The protein catabolic state of cirrhosis is associated with severe growth hormone (GH) resistance, with low levels of insulin-like growth factor (IGF)-I and its major binding protein (IGFBP)-3 . GH therapy in cirrhosis have been shown to improve nitrogen economy and to improve the GH resistance in a small pilot study. Also, GH therapy of short duration has shown to increase IGF1 levels, IGFBP-3 levels in patients of cirrhosis . GH therapy has also shown to improve liver regeneration and protein synthesis after hepatectomy in patients of HCC with cirrhosis . However there is scarcity of data on clinical impact of long term administration of GH therapy in patients of cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

Decompensated Cirrhosis of liver.

Exclusion Criteria:

* Acute on chronic liver failure
* Spleen diameter of larger than 180 mm
* Diagnosis of concomitant hepatocellular carcinoma or other active malignancy
* Upper gastrointestinal bleed due to portal hypertension in the previous 7 days
* Recent episode of portal vein thrombosis
* Severe renal dysfunction creatinine (>1.5mg/dl)
* Severe cardiac dysfunction
* Uncontrolled diabetes or diabetic retinopathy
* Acute infection or disseminate intravascular coagulation
* Active alcohol abuse in last 3months
* Known hypersensitivity to G-CSF and GH
* Human immunodeficiency virus seropositivity
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Transplant free survival | 1 year
  Survival at 1 year from the onset of therapy

SECONDARY OUTCOMES:
haematopoietic stem cell mobilization | 1 year
  Mobilisation of CD34+ cells in peripheral blood
safety as measured by adverse effects of G-CSF, GH and combination in cirrhosis of liver | 1 year
  Adverse effects of G-CSF, GH and combination in cirrhosis of liver
Clinical/biochemical improvement in liver function profile | 1 year
  Improvement in prognostic scores - MELD score, and Child score

CONTACTS AND LOCATIONS:
Overall Officials: Virendra Singh, MD;DM, Principal Investigator — Professor of Hepatology,PGIMER,Chandigarh
Locations (2):
- India (2):
  - Dept. of Hepatology, PGIMER, Chandigarh, Chandigarh
  - Department of Hepatology,Postgraduate Institute of Medical Education and Research, Chandigarh

REFERENCES:
- [Derived] Kaur A, Verma N, Singh B, Kumar A, Kumari S, De A, Sharma RR, Singh V. Quantitative liver SPECT/CT is a novel tool to assess liver function, prognosis, and response to treatment in cirrhosis. Front Med (Lausanne). 2023 Mar 22;10:1118531. doi: 10.3389/fmed.2023.1118531. eCollection 2023. PMID 37035316
- [Derived] Verma N, Kaur A, Sharma R, Bhalla A, Sharma N, De A, Singh V. Outcomes after multiple courses of granulocyte colony-stimulating factor and growth hormone in decompensated cirrhosis: A randomized trial. Hepatology. 2018 Oct;68(4):1559-1573. doi: 10.1002/hep.29763. Epub 2018 Jul 25. PMID 29278428